CLINICAL TRIAL: NCT07136441
Title: Sciatic Nerve Stiffness Using Two-Sequences of Lower Limb Neurodynamic Testing: A Shear Wave Elastography Study
Status: Recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Manar Fawzy Mohamed, Principal Investigator, Cairo University
Other Study IDs: P.T.REC/012/005897
Record Dates: First submitted 2025-08-05; First posted 2025-08-22 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Sciatic Nerve

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A (Low Back Pain with Sciatica): Thirty patients with low back pain with sciatica aged 25-40 years with unilateral leg pain for 3-12 months, lumbar disc herniation (L4-5) confirmed by MRI, and positive straight leg raising test. Participants will receive sciatic nerve tension tests using both proximal-to-distal and distal-to-proximal sequences with shear wave elastography assessment.
  Interventions: Diagnostic Test: Lower Limb Neurodynamic Test (LLNT) with Shear Wave Elastography
- Group B (Control Group): Thirty healthy control participants aged 25-40 years, free from symptoms of nerve irritation or compression, with normal neurological examination findings including normal reflexes, sensation, negative straight leg raising test, and normal motor strength. Participants will receive the same sciatic nerve tension tests in both sequences.
  Interventions: Diagnostic Test: Lower Limb Neurodynamic Test (LLNT) with Shear Wave Elastography

INTERVENTIONS:
Diagnostic Test: Lower Limb Neurodynamic Test (LLNT) with Shear Wave Elastography — Participants underwent sciatic nerve stiffness assessment using shear wave elastography during two distinct sequences of the lower limb neurodynamic test. Each participant received:
  Proximal-to-distal sequence: Starting with hip flexion, followed by knee extension, then ankle dorsiflexion with toe extension.
  Distal-to-proximal sequence: Starting with ankle dorsiflexion and toe extension, followed by knee extension, then hip flexion.
  Other Names: Two-Sequence Neurodynamic Testing

SUMMARY:
The purposes of the study are:

1. To measure differences in Sciatic nerve (SN) stiffness using shear-wave elastography (SWE) during two movement sequences of the lower limb neurodynamic test (LLNT) in low back pain with sciatica.
2. To measure differences in Sciatic nerve stiffness using shear-wave elastography during two movement sequences of the lower limb neurodynamic test in control group.
3. To compare difference in Sciatic nerve stiffness using shear-wave elastography during two movement sequences of the lower limb neurodynamic test between low back pain patients with sciatica and control group.

DETAILED DESCRIPTION:
As peripheral nerves can exhibit regional variations in their anatomy and mechanical properties, investigating the response of different nerve segments to different loading patterns based on the order of joint movement will provide a better understanding of nerve biomechanics during neurodynamic testing.

This may help optimize the lower limb neurodynamic test (LLNT) application for different pathological situations and potentially increase its diagnostic capacity to detect localized alterations in a specific nerve segment such as sciatica.

Ultrasonography does not have the sensitivity required to detect all forms of peripheral nerve disorders and fails to provide information about nerve mechanical properties such as stiffness.

By using neurodynamic sequencing, clinicians may direct neural stress toward targeted areas suspected of involvement and, at the same time, perform the test with reduced load on more remote nerve segments. The ability to modify neural load distribution during the LLNT could play an interesting role in differential diagnosis, when symptoms present similar characteristics but have different regional origin.

There is a gap in the literature concerning the measurement of (SWV) of sciatic nerve during LLNT proximal (LLNT-PROX) to distal and from distal (LLNT_DIST) to proximal sequences of LLNT.

ELIGIBILITY:
Inclusion Criteria:

* Thirty participants ranging in age from 25 to 40 years from both genders with a diagnosis of low back pain with radiating leg pain and thirty control group.
* The main symptoms are low back pain with unilateral leg pain(sciatica) for 3-12 months for group A.
* Patients with lumbar disc herniation (L4-5) with diagnostic imaging as MRI for group A.
* Positive straight leg raising are considered for inclusion in the study for group A.
* Control group must be free from any symptoms of nerve irritation or compression, with normal neurological examination findings, including reflexes, sensation, negative straight leg raising and motor strength.

Exclusion Criteria:

* Diabetes mellitus.
* Any type of polyneuropathy
* Trauma of lumbar spine
* Previous history of back surgery
* Piriformis syndrome.
* Participants with conditions that reduce image quality on US imaging (thick gluteal subcutaneous fat tissue.
* Hip joint prosthesis.
* Professional athletes (Neto et al., 2024).
* Skin infection

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Sixty subjects of both genders will be participated in this study. Their age will range between 25 to 40 years. They will receive verbal and written explanations for this study. If they decide to participate in this study, they will sign the consent form. The sample will be selected from the faculty of physical therapy outpatient clinics and at El kasr Elainy.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Shear Wave Velocity (SWV) measured in meters per second (m/s) | 20 minutes, During a single assessment session at baseline
  Quantitative measurement of sciatic nerve stiffness during two different movement sequences of the Lower Limb Neurodynamic Test (LLNT). Higher SWV values indicate increased nerve stiffness.

CONTACTS AND LOCATIONS:
Overall Officials: Eman Ahmed Abd Elmoez, PhD, Study Chair — Professor, Cairo university; Najlaa Fathi Ewais, PhD, Study Director — Assistant Professor, Cairo university; Ebtisam Abdelkareem Ali, PhD, Study Director — Lecturer, Cairo university; Hatem Mohamed El-Azizi, PhD, Study Director — Professor, Cairo university
Locations (1):
- Cairo University, Giza, Egypt